CLINICAL TRIAL: NCT00343655
Title: A Randomized Clinical Trial Of Atorvastatin 10 Mg And 80 Mg In The Reversal Of Or Stabilization Of Carotid Atheroma Lipid Pool
Brief Title: Evaluation of Atorvastatin Treatment on Carotid Plaque.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated on June 22, 2007 for inability to enroll patients within an appropriate timeframe. There were no efficacy/safety concerns.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581152
Record Dates: First submitted 2006-06-20; First posted 2006-06-23 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases
Keywords: Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The purpose of the study is to evaluate the effect of 18 months treatment with atorvastatin 80mg or atorvastatin 10mg on the carotid vessel plaque morphology, in particular, the effect on evident necrotic lipid rich core of the plaque in patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with measurable carotid plaque with lipid and are eligible for statin therapy.

Exclusion Criteria:

* Subjects at higher risk for cardiovascular disease with a screen LDL-cholesterol greater than 120 mg/dL,
* Subjects currently on high dose statin, and
* Subjects with contraindications for MRI or statin therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in lipid pool volume from baseline to 18 months in response to atorvastatin 80mg.
Comparison of effect of atorvastatin 80mg versus 10mg

SECONDARY OUTCOMES:
Correlation of MRI measure of carotid morphology with cIMT measured by B-mode US.
Correlation of MRI measure of carotid morphology with DS-CT measure of coronary morphology.
Correlation of biomarkers to carotid changes.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Boston, Massachusetts, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581152&StudyName=Evaluation%20of%20Atorvastatin%20treatment%20on%20carotid%20plaque.%20